CLINICAL TRIAL: NCT01118988
Title: Peer Mentorship: An Intervention To Promote Effective Pain Self-Management In Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lonnie Zeltzer, Distinguished Professor of Pediatrics, Anesthesiology, Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HD057421-01A2 (NIH)
Record Dates: First submitted 2010-04-27; First posted 2010-05-07 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Irritable Bowel Syndrome (IBS); Functional Abdominal Pain; Fibromyalgia; Complex Regional Pain Syndrome (CRPS); Myofacial Pain; Chronic Daily Headaches; Migraine Headaches; Chronic Pain
Keywords: Peer Support; Social Support; Chronic Pain; Behavioral Interventions for Pain; Adolescents; Children; Pediatric; Mentorship; Complementary and Alternative Medicine; CAM; Pain; Pain Management; Behavioral
MeSH Terms: conditions — Irritable Bowel Syndrome; Fibromyalgia; Complex Regional Pain Syndromes; Facial Pain; Headache Disorders; Migraine Disorders; Chronic Pain; Pain; Agnosia; Behavior | interventions — Palliative Care; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mentorship (Experimental): Subjects randomly assigned to this arm received the specified "Mentorship Intervention"
  Interventions: Behavioral: Mentorship
- Control (No Intervention): Subjects randomly assigned to this control group receive treatment as usual (TAU).
- Mentors (No Intervention): Subjects recruited to the "Mentor" arm of the study are UCLA Pediatric Pain Program patients between the ages of 14 and 18. These mentors are identified by the Principal Investigator as children who have not necessarily eliminated pain, but have learned how to cope with pain and maintain appropriate functioning in daily life. Mentors undergo an in depth training from doctoral level psychologists who are members of the research team. Mentors present pain coping information developed by the research team, provide support, and encourage mentees to attend pain management therapies. They are also monitored by doctoral level psychologists throughout the duration of the study to ensure safety and appropriate contact with mentees via telephone.

INTERVENTIONS:
Behavioral: Mentorship — Subjects in this condition receive 10 sessions over 8 weeks (2 sessions for the first 2 weeks, 1 session per week for the remaining 6 weeks) with a mentor presenting information on pain self-management and coping techniques, as well as discussing concerns and feelings with the subject receiving the intervention. Information is presented on slides via internet connected home computer. Mentor-mentee interaction is conducted via telephone on a conference call line with a doctoral level psychologist monitoring call for safety of all parties.
  Other Names: support; education
  Arms: Mentorship

SUMMARY:
This protocol matches child subjects with peer mentors of similar age who have learned to function successfully with a chronic pain disorder. The trained mentors will present information to the subjects in a supervised and monitored interaction via telephone and computer for 2 months and encourage participation in skill-building programs. Children will be tested for improvement in pain and functioning at 2 months and again at 4 months to see if improvements persist. The investigators hypothesize that children who received peer mentor support will show more improvement in pain and functioning at 2 and 4 months into treatment than those in a control group who do not receive mentor support.

DETAILED DESCRIPTION:
Background:

Chronic intractable non-malignant pain, including such functional disorders as irritable bowel syndrome is now recognized as a significant problem in children and adolescents, with potential long-term impact on the child's physical, social, and academic functioning, as well as on the family as a whole. A recent study of more than 5000 Dutch school children under 18 found that more than 25% reported suffering recurrent or continuous pain for more than 3 months, with the prevalence increasing with age; and a survey of 735 German children aged 10-18 using a modified version of the same instrument found the same for 45.5%. The most common types of pain in these two studies were headache, abdominal pain, limb pain, and back pain. This data would appear to confirm earlier estimates that recurrent headache, including migraine, occurs in 11% to 26% of children ages 7-15; recurrent abdominal pain in 10-15% and recurrent limb pain in 4-18% in children ages 7-15. Many such children apparently continue to function effectively, attending school and continuing normal activities, with medical intervention only for acute episodes. A smaller, but significant, number, however, find themselves unable to self-manage their pain. They become patients with chronic pain and disability, falling into a cyclical pattern of pain, impaired functioning in physical, school, social, and even family and self-care domains, "doctor-seeking" and over-utilization of medications, and psychosocial distress, including anxiety and depression.

Functional impairment, particularly in academic work and social participation, is likely to have long-term effects on the individual's quality of life, even aside from the possibility that pain and physical limitations may persist into adulthood. Several well-designed studies using quantitative measures have provided evidence that impaired functioning in children with chronic pain is strongly associated with psychosocial distress and with lower quality of life. In particular, children with unexplained chronic pain, pain not associated with an organic diagnosis, often report significant dysfunctions in normal activities, such as schoolwork, sleep, family activities, and athletic activities. But, although impaired functioning is a major factor in lower quality of life for children with chronic pain, we still know relatively little about the prevalence and severity of functional impairment, why some children experience more limitations than others, and which treatment interventions are the most effective in improving function.

The available evidence also indicates that children show different levels of adjustment to chronic pain over time. Chronic idiopathic musculoskeletal pain has been shown to persist in 59% of cases for as long as nine years; in this study, the authors found the children to have pain and disability levels comparable to children with juvenile chronic arthritis, but lower levels of psychosocial functioning. Hunfeld, Perquin, and colleagues in Rotterdam have traced the persistence of chronic benign pain in 30-45% of cases for up to two years and three years, with no increase in intensity or frequency. In the latter study, open-ended interviews elicited information about functioning and coping skills, and identified continuing problems with physical activity, mental concentration, social interaction, and psychological stress (becoming "moody"), particularly when the pain was severe. The researchers found, however, that several children had developed their own strategies to maximize functionality despite the continuing pain: "…pain had become part of the daily lives of several adolescents, who structured their activities and sleeping hours to prevent aggravation of pain". A recent cluster analysis of 117 children with chronic pain divided them into three groups on the basis of a set of psychosocial and behavioral measures: those who were highly distressed and disabled; those who showed low levels of distress and disability; and those who showed only moderate levels of distress and disability, but whose family environment scored low on cohesion.

Although several factors may account for children's differential ability to function and to adjust to persistent chronic pain, the child's sense of self-competence has been identified as a key variable in recent literature. Claar and colleagues, for example, found that in adolescents and young adults with irritable bowel syndrome, the relationship between pain and functional disability was moderated by the individual's sense of academic, social, and athletic competence. The concept of self-competence (a general sense of mastery) overlaps with that of self-efficacy (a task-specific sense of mastery), developed by Albert Bandura in the late 1970s and early 1980s 18. The concept of self-efficacy suggests an explanation for the relationship between coping skills, perceived ability to cope, and reduction in physical and psychological disability. Bandura argued that a sense of self-efficacy enables the individual to persist even with a task of great difficulty until it is mastered, to reject negative thoughts and to "bring cognitive or cerebral productions into being" that will assist in achieving the goal.

To summarize briefly, impaired functioning in all domains is a major and potentially a long-term problem for children with recurrent or chronic pain and their families, which are a significant segment of the American population. Children show significant variations in their ability to cope with pain and continue to function, and some children learn better functioning over time. The child's own sense of self-competence, or task-specific self-efficacy, is one important factor which may reinforce or moderate the child's functioning. Functional disability is clearly associated with psychosocial distress. But these factors are also mutually reinforcing; while children with more psychosocial distress may have more problems functioning with pain, certainly children who experience pain and attendant functional problems are likely to react with anxiety and/or depression.

Current Therapeutic Interventions: When chronic pain can not be fully alleviated, the optimal goal is for the patient to learn effective ways to continue functioning and to self-manage pain; several therapeutic programs have been developed, based on theories of health behavior change, to assist the patient in this process. The earliest of these, the operant learning model developed by Wilbert Fordyce and colleagues in the late 1970s, demonstrated that individuals could be induced to alter their behavior - specifically, to engage in active exercise and limit dependence on medication - in response to social and other forms of positive reinforcement. Fordyce's program proved helpful to many patients, but was criticized for its determinist emphasis on observable behavior and disregard of the fact that patients are "active information processors", and that their behavior is not merely a response to learned cues but shaped by cognitive processes, such as expectations of increasing pain or anxieties about physiological harm.

The revised therapeutic programs that developed in response to these criticisms drew on overlapping models linking health beliefs to health behavior and to self-efficacy as described by Bandura. These new models rely on an expectancy-value theory of behavior; that behavioral change is not a simple learned response to reinforcement, but that learning is influenced by the individual's cognitive belief (expectancy) that s/he will be able to change functioning with positive consequences (self-efficacy) and by his/her expectations (values) of the potential benefits of and barriers to behavioral change. Thus the new therapeutic programs, the most well-known and widely practiced of which is cognitive-behavioral therapy (CBT), seek to mediate behavioral change through cognitive relearning. The cognitive behavioral therapist uses a number of methods -- including education about pain, verbal reinforcement for positive cognitions and actions, biofeedback, group therapy allowing patients to observe and learn from each other, and teaching of cognitive tools to repress negative thoughts -- to help the patient develop positive expectations of behavior change, minimize negative expectations, and internalize the conviction of his/her own ability to overcome barriers and effectively self-manage pain In effect, the patient becomes the agent of change.

CBT has been shown to be effective in controlled trials of treatment pain in cancer patients; of chronic low-back pain; of osteoarthritic knee pain; of sickle cell disease; of pediatric migraine; and of recurrent abdominal pain in children. CBT with family involvement has been found to be an effective intervention for adolescents with chronic pain and chronic fatigue 31-33. Flor, Fydrich, and Turk's 1992 analysis of 65 studies of multidisciplinary treatments for chronic low back pain in adults, covering a number of variants of cognitive, behavioral, and coping skills training packages, noted that many of the studies were "marginal" in quality, but nevertheless demonstrated that these methods were superior to no treatment and to single-modality treatment -- medical or physical therapy -- in decreasing pain and impairment, improving mood, promoting return to work, and decreasing health services utilization. "Even at follow up, patients...are functioning better than 75%" of control groups; the findings of efficacy are "quite impressive". A recent systematic review of behavioral treatment for low back pain again found only six studies "of high quality". The authors nevertheless thought the evidence strong that behavioral therapy had at least "a moderate positive effect" on pain intensity and "small positive effects" on functional status; but they noted that "it is still unknown what type of patients benefit most" from behavioral therapies.

A well-designed intervention, it appears, is not enough: not all patients will benefit from CBT. As Dennis Turk, the leading exponent of CBT, has stated, patient motivation is at least one of the critical factors in successful outcomes of this therapeutic model. Jensen and colleagues have recently proposed a cogent general model that integrates the varied theoretical approaches to describe a dynamic process that pivots on this concept of motivation, or readiness to change. An individual's readiness to change, they argue, is essential to his/her ability to learn successful pain self-management through new behaviors; and readiness is a dynamic function of 1) his/her perceived importance of the change (beliefs of the costs and benefits of change, past experience with change (learning history), and current contingencies (availability of social and material support) and 2) his/her self-efficacy beliefs (personal experience, modeling provided by others, verbal persuasion, and perceived barriers). They suggest some clinical approaches for enhancing readiness and promoting change, including encouragement to practice self-management; allowing the patient to observe other pain patients practice self-management; support of positive beliefs and non-judgmental non-support of negative beliefs; and development of a plan to address real or perceived barriers; and they call for research into interventions along these lines to enhance motivation.

Another formulation recently proposed by Sharp stresses the patient's cognitive activity in appraising and evaluating his or her pain, and its ongoing and interactive effects on mood, behavior, and somatic focus. The patient's initial response to the pain is a function of cultural beliefs, learning history, and current contingencies, he argues, but then is continually reinterpreted with ongoing events. In particular, anxiety about recurrent pain and avoidance of activity that might cause pain will help to perpetuate the patient's hypervigilance for signs of recurring pain (as described by Eccleston and Crombez) and his/her perceived inability to manage the pain. Moreover, Sharp contends that this attitude of "learned helplessness" may be perpetuated by physicians who have failed to offer helpful treatment or even to confirm the physical reality of the patient's suffering. "That is, patients could start to believe that 'nothing has worked so far so why would any future treatment help?" A patient who has reached this point is likely to have a negative assessment both of the benefits of pain self-management and of his/her own ability or self-efficacy to learn these skills, and will therefore show a lack of readiness to change.

In this study, we will consider adolescent pain patients and whether a new type of innovation can promote their readiness to change and to learn pain self-management skills, that will promote positive outcomes in pain reduction and improved functioning.

Findings from our Current Research: Our interdisciplinary group, comprised of researchers from anthropology, history, pediatrics, psychology, and sociology, has collected quantitative and interview data on 74 adolescent children presenting between 2003 and 2006 to the Pediatric Pain, Pediatric Gastroenterology, and Pediatric Neurology Clinics with recurrent or persistent pain. We have completed preliminary analysis of the qualitative data for a subset of 37 (28 girls and 9 boys, average age 13.97) for whom intake and six-month follow-up data was obtained. These children reported suffering pain for periods ranging from one month to "all my life": the average computed duration was 53.6 months, or about 4.5 years. All of them had seen at least one physician prior to referral to UCLA and the majority had seen three or more.

The children's levels of functioning varied considerably on the quantitative measures, but the evidence from the long, semi-structured interviews (conducted prior to the first Clinic appointment and at 6 months) shows that virtually all were distressed by some level of impairment. Those who had had pain for several years reported that pain had become part of daily life and that they adjusted their lives around it: Many of the children also stated that their unexplained chronic pain, which a series of doctors had not been able to diagnose, had given them a sense of isolation and difference from others, and a sense of powerlessness, that contributed to their distress:

Those children seen in the Pediatric Pain Clinic (28, or 76% of the 37) were given recommendations to choose one or more of a list of complementary and alternative medicine (CAM) providers who work with the clinic; these include several who teach pain self-management skills, including a physical therapist, yoga therapist, biofeedback trainer, and guided imagery/hypnotherapist. These recommendations were made in addition to those for tests, changes in medication or other therapies. Children seen in the GI or Neuro Clinic might be given a recommendation for PT or another CAM treatment, but it was not a standardized part of the treatment plan. At the follow-up interview, the children were asked whether their pain and functioning had improved, and also to talk about their participation in any of the CAM therapies:

Better, pain improved or resolved by medication change - 8; 22%

Better, participation in active CAM had helped - 8; 22%

Better, medication change and participation in an active CAM therapy - 4; 11%

Same, meds had not helped, no interest in CAM - 6; 16%

Same, meds had not helped, CAM not tried because not recommended or because of reimbursement issues - 5; 13%

Same, meds had not helped, child tried CAM but did not persist - 2; 6%

Worse, meds had not helped, no interest in CAM - 1; 3%

Worse, meds had not helped, CAM too expensive - 1; 3%

Worse, meds had not helped, child tried CAM but did not persist - 1; 3%

Worse for other reasons (intervening surgery had increased pain) - 1; 3%

These findings are not presented as supportive evidence of the benefits of CAM therapy. Rather, they indicate, that, in this group of children, aside from a small group helped by a medication change and one outlier case, those who were self-motivated to participate in a therapy that taught them active self-management consistently reported better outcomes than those who were not self-motivated or who were unable to do so.

Why did 16 of the children choose not to participate or persist in participating in recommended CAM therapy? One possible explanation is that they lacked confidence that a new therapy will work when many others have failed to work and believed that their pain was a different and intractable problem that doctors did not know how to treat and that they could not manage themselves. Another is that they were not given the opportunity to observe others; were not given sufficient reinforcement from family or other significant contacts for participation; and were not helped to overcome any perceived barriers to access.

On the basis of this preliminary data, considered in the light of current theoretical models, we propose the following hypotheses:

* Adolescents who participate actively in learning a pain-management skill will show more improvement in pain and functioning at 2 and 4 months than those who do not.
* Adolescents who lack peer support for learning a pain management skill will not follow through with learning such a skill without further reinforcement, even if recommended as part of a treatment plan.
* Adolescents may be helped to adhere to treatments that involve learning a pain management skill which will improve their pain and functioning by talking to others who have learned such a skill; by receiving ongoing positive reinforcement; and by being helped to overcome perceived barriers.

We propose to test our hypotheses through a trial of a peer mentorship intervention, using trained adolescents who have successfully learned pain management skills as mentors. The mentor will help to relieve the child's sense of isolation and difference by relating their similar experiences, provide models of successful skill learning and reinforce the mentored subject's participation in skill learning activities.

ELIGIBILITY:
Mentors

Inclusion criteria:

* between the ages of 14 and 18
* any patient who has been successfully treated in the UCLA Pediatric Pain Program
* access to telephone
* access to internet enabled computer

Exclusion criteria

* younger than 14
* older than 18
* new patient
* no access to telephone
* no access to internet enabled computer

Mentees and controls:

Inclusion Criteria:

* chronic pain diagnosis
* between the ages of 12 and 17
* access to telephone
* access to internet enabled computer
* new to UCLA Pediatric Pain Clinic
* plans to utilize program CAM therapies

Exclusion Criteria:

* already utilizing UCLA Pediatric Pain Program CAM therapies
* unable to read, speak, or understand english
* younger than 12 or older than 17
* no access to telephone
* no access to internet enabled computer
* not new patient to UCLA Pediatric Pain Clinic
* does not plan to utilize program CAM therapies

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lonnie K. Zeltzer, MD, Principal Investigator — UCLA Department of Pediatrics
Locations (1):
- UCLA Pediatric Pain Management Clinic, Los Angeles, California, United States

REFERENCES:
- [Derived] Allen LB, Tsao JC, Hayes LP, Zeltzer LK. Peer mentorship to promote effective pain management in adolescents: study protocol for a randomised controlled trial. Trials. 2011 May 22;12:132. doi: 10.1186/1745-6215-12-132. PMID 21600053

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mentorship | Control | Mentors
Started | 16 | 4 | 7
Completed | 11 | 3 | 3
Not Completed | 5 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mentorship | Control | Mentors | Total
Number analyzed (Participants) | 16 | 4 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.44 (1.71) | 15.35 (0.31) | 16.88 (1.49) | 15.80 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 6 | 20
  Male | 5 | 1 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 9 | 3 | 5 | 17
  Unknown or Not Reported | 4 | 1 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 8 | 3 | 5 | 16
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 5 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Physician Recommended CAM Therapies
Description: This measure tracks the attendance of CAM therapies recommended by the subjects' pain specialist physician.
Time Frame: post intervention (week 8)
Population: One participant in the Mentorship group did not do the weekly CAM therapy tracking and is thus not included in the results for this measure.
Measure: Mean (Standard Deviation); unit: Visits to CAM therapists per week
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 10 | 3
Visits to CAM therapists per week | 1.34 (0.64) | 2.23 (1.19)

2. Secondary Outcome: Body Map and Pain Assessment
Description: visual depiction of body pain and associated pain ratings over certain periods of time and conditional situations
  Range: 0-19 body areas
Time Frame: 2 months
Population: Not all participants who completed the intervention completed this measure, so the numbers reported herein are lower than those reported in Participant Flow.
Measure: Mean (Standard Deviation); unit: Number of painful body areas
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 9 | 2
Number of painful body areas | 7.56 (6.69) | 8.50 (6.36)

3. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: assessment of sleep quality
  Range: 0-21; higher scores = lower sleep quality
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 6 | 2
units on a scale | 9.67 (4.13) | 7.50 (2.12)

4. Secondary Outcome: Child Symptom Inventory (CSI)
Description: Assement of somatic symptom complaints
  24 items, range 0-96, higher score = more somatic symptoms
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale | 33.64 (17.04) | 26.00 (2.83)

5. Secondary Outcome: Child Anxiety Sensitivity Inventory (CASI) - Child Report
Description: Assessment of child's anxiety sensitivity
  18 items, range 18-54, higher scores = more anxiety sensitivity
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale | 29.38 (5.73) | 24.50 (6.36)

6. Secondary Outcome: Health Belief Scale (HBS) Short Version - Child Report
Description: Number of treatment modalities rated 1-4 by participants on the HBS questionnaire, which asked participants to rate how much they think each of 16 listed treatment modalities would help with pain (1=Completely, 2=A lot, 3=Some, 4=A little, 5=Not at all).
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of treatments
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 9 | 2
Number of treatments | 10.89 (3.14) | 10.00 (0.00)

7. Secondary Outcome: Emotion Regulation Questionnaire (ERQ) - Child Answer
Description: assessment of child emotion regulation
  Reappraisal subscale: 6 items, range 6-30, higher scores = higher use of reappraisal Suppression subscale: 4 items, range: 4-20, higher scores = higher use of suppression
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale
  Reappraisal | 23.63 (4.96) | 25.00 (1.41)
  Suppression | 9.38 (3.02) | 9.00 (0.00)

8. Secondary Outcome: Emotion Expression Scale for Children (EESC)
Description: assess child emotional expression/emotion regulation
  Poor Awareness subscale, 8 items, range: 8-40; higher scores = poorer emotional awareness Expressive Reluctance subscale, 8 items, range: 8-40; higher scores = more expressive reluctance
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale
  Poor Awareness | 16.88 (4.97) | 10.0 (1.41)
  Expressive Reluctance | 16.75 (6.92) | 12.0 (1.41)

9. Secondary Outcome: Functional Disability Inventory (FDI)
Description: assesses functional disability for daily tasks
  Range: 0-60; higher scores mean greater functional disability.
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale | 25.88 (16.57) | 18.00 (8.49)

10. Secondary Outcome: Revised Child Anxiety and Depression Scale (RCADS) Child Report
Description: assess levels of symptoms for anxiety disorders and depression
  Range: 0-141; Higher scores mean higher symptom level of anxiety and depression
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale | 39.44 (20.32) | 20.00 (12.73)

11. Secondary Outcome: Beck Depression Inventory 2 (BDI-2) #18
Description: assesses suicidal ideation and intent
  Number reported is number of participants who reported any level of suicidal ideation or intent at any time and who were followed with the study's emergency protocol to ensure that such participants are not a threat to self or others, and that he/she was under the appropriate mental health care.
Time Frame: baseline, weekly weeks 1-8, 2 months, 4 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 9 | 2
participants | 1 | 0

12. Secondary Outcome: Child Health Questionnaire - Child Report (CHQ)
Description: detailed questionnaire about health, daily activites, pain, behavior, family health, self-esteem
  Subscales (for all subscales, higher scores = better health):
  Behavior - 16 items, averaged, range 1-5 Bodily Pain and Discomfort - 2 items, averaged, range 1-6 Change in Health - 1 item, range 1-5 Family Activities - 6 items, averaged, range 1-5 Family Cohesion - 1 item, range 1-5 Global Health - 1 item, range 1-5 Global Behavior - 1 item, range 1-5 General Health - 12 items, averaged, range 1-5 Mental Health - 16 items, averaged, range 1-5 Physical Functioning - 9 items, averaged, range 1-4 Role/Social Limitations Behavioral - 3 items, range 1-4 Role/Social Limitations Emotional - 3 items, range 1-4 Role/Social Limitations Physical - 3 items, range 1-4 Self-Esteem - 14 items, range 1-5
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale
  Behavior Sub-Scale | 4.12 (.54) | 4.66 (.07)
  Bodily Pain and Discomfort Sub-Scale | 1.69 (.59) | 2.50 (0.00)
  Change in Health Item Sub-Scale | 2.71 (1.38) | 2.50 (.71)
  Family Activities Sub-Scale | 3.26 (.99) | 3.63 (.05)
  Family Cohesion Item Sub-Scale | 4.17 (.90) | 3.90 (.71)
  Global Health Item Sub-Scale | 2.33 (1.30) | 3.30 (1.56)
  Global Behavior Item Sub-Scale | 4.20 (1.05) | 4.70 (.42)
  General Health Perceptions Sub-Scale | 2.50 (.84) | 2.61 (.13)
  Mental Health Sub-Scale | 3.67 (.48) | 3.81 (.35)
  Physical Functioning Sub-Scale | 2.87 (.86) | 3.67 (.16)
  Role/Social Limitations due to Behavioral Difficul | 3.42 (1.05) | 4.00 (0.00)
  Role/Social Limitations due to Emotional Difficult | 2.96 (1.25) | 3.50 (.71)
  Role/Social Limitations due to Physical Health | 2.13 (1.25) | 3.17 (.24)
  Self-Esteem Sub-Scale | 3.64 (.76) | 3.58 (.92)

13. Secondary Outcome: Positive and Negative Affect Scale (PANAS)
Description: assesses extent to which children have felt a number of positive and negative affects
  Positive Affect subscale, 12 items, range: 12-60, higher score = more positive affect Negative Affect subscale, 15 items, range: 15-75, higher score = more negative affect
Time Frame: 2 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentorship | Control
Number analyzed (Participants) | 8 | 2
units on a scale
  Positive Affect | 38.95 (9.60) | 32.00 (8.49)
  Negative Affect | 29.38 (8.45) | 24.00 (8.49)

ADVERSE EVENTS:
Arm/Group | Mentorship | Control | Mentors
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/16 | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No